CLINICAL TRIAL: NCT02574962
Title: Pilot Study of Acthar® Gel in Chronic Inflammatory Demyelinating Neuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Mamatha Pasnoor, MD (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Mamatha Pasnoor, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002770
Record Dates: First submitted 2015-08-30; First posted 2015-10-14 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acthar® Gel (Experimental): For the first two weeks participants will receive 1 mL of study drug subcutaneously every other day. After that, participants will received 1 mL of study drug twice a week for up to 6 months.
  Interventions: Drug: H.P. Acthar® Gel

INTERVENTIONS:
Drug: H.P. Acthar® Gel
  Other Names: Acthar® Gel; repository corticotropin injection

SUMMARY:
The purpose of this pilot study is to assess the safety and efficacy of Acthar® Gel in Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) patients.

ELIGIBILITY:
Inclusion Criteria:

* CIDP diagnosed according to the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) criteria 2010
* Age > 18 years
* Able to give written informed consent
* Patient's signs and symptoms should not be better explained by another disease process
* Patients can be on prednisone as long as there has been no dose change for 4 weeks from baseline
* Patients can be on following drugs as long as there has been no change for 60 days from baseline visit including azathioprine, cyclosporine, cyclophosphamide, mycophenolate mofetil, intravenous immunoglobulin (IVIg) or other immunosuppressive drugs
* INCAT score greater than or equal to 2

Exclusion Criteria:

* Presence of any other causes of polyneuropathy or multifocal motor neuropathy, which in the opinion of the investigator is the major contributor to the numbness and weakness.
* Other neurologic or orthopedic condition causing weakness
* Treatment with plasma exchange (PLEX) within the last 30 days from baseline
* Participation in another trial within the last 30 days from baseline or two ½ life of the drug being studied.
* Latent tuberculosis or active infection
* Contraindication per Acthar® Gel prescribing information scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history or presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction.
* History of prior sensitivity to Acthar® Gel or other porcine products
* Previous or present Infection with hepatitis C and hepatitis B
* Pregnancy or nursing mothers.
* Female subjects of childbearing potential either not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study, or not sexually abstinent for the entire duration of the study, or not surgically sterile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events | 28 Weeks
  Count of adverse events experienced by study participants.

SECONDARY OUTCOMES:
Efficacy of study drug | Change from Baseline to 28 Weeks
  Measured using the Inflammatory Neuropathy Cause and Treatment (INCAT) score. The INCAT scale has upper and lower extremity components (maximum of 5 points for upper (arm disability) and maximum of 5 points for lower (leg disability) that add up to a maximum of 10-points. A score of 0 indicates no problems. A score of 10 indicates person is severely incapacitated.

OTHER OUTCOMES:
Maximum Grip Strength | 28 weeks
  Measured by the amount of force a person uses to squeeze around a dynamometer.
Manual Muscle Testing (MMT) | 28 Weeks
  Measure based on the Medical Research Council (MRC) sum score (strength score combined for 12 specified muscle groups) on MMT.
Rasch-built Overall Disability Scale (R-ODS) | 28 Weeks
  The R-ODS is a questionnaire that rates a person's ability to perform 24 daily activities such as eating, using the toilet, taking a shower, dressing, walking, dancing, running, or standing. Scores range from 0-48 with 0 meaning they cannot perform any of the tasks and 48 meaning they can perform all of the tasks without any difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Mamatha Pasnoor, MD, Principal Investigator — University of Kansas Medical Center
Locations (5):
- United States (5):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wesley Neurology Group, Memphis, Tennessee
  - University of Vermont, Burlington, Vermont